CLINICAL TRIAL: NCT02700074
Title: ACE (Autism Center of Excellence): Brain Mechanisms for Language Processing in Adolescents With Autism Spectrum Disorder
Brief Title: Brain Mechanisms for Language Processing in Adolescents With Autism Spectrum Disorder
Acronym: BSL
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Massachusetts General Hospital (Other); Northeastern University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Helen B. Tager-Flusberg, Professor, Boston University
Other Study IDs: 3077E; P50DC013027 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Minimally Verbal: Minimally verbal adolescents with Autism Spectrum Disorder
  Interventions: Other: No Intervention
- Verbal Impaired: Language impaired adolescents with ASD
  Interventions: Other: No Intervention
- Verbal Normal: Language normal adolescents with ASD
  Interventions: Other: No Intervention
- Typically Developing: Typically developing adolescent controls
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Intervention is not a part of this study.

SUMMARY:
The main goal of our study is to find out why some people with Autism Spectrum Disorder (ASD) do not develop verbal abilities or remain minimally-verbal throughout adolescence and adulthood. Current research focuses on investigating brain differences related to processing sounds and initiating speech in adolescents and young adults with ASD varying in language skills, compared to adolescents who do not have ASD, in order to clarify whether atypical processes of auditory perception, perceptual organization and/or neural oscillation patterns may explain why some individuals with ASD fail to acquire functional speech.

DETAILED DESCRIPTION:
About 30% of children with Autism Spectrum Disorder (ASD) fail to acquire spoken language. This group of children has been seriously neglected in research conducted over the past 2 decades. Little is known about them, in part because the field lacks the tools to assess them, and they often pose significant behavioral challenges that preclude their participation in research studies. Among the ~70% individuals with ASD who have spoken language skills, about 50% are language impaired; the remaining group have normal language scores on standardized tests. Thus, there is enormous heterogeneity in verbal abilities in ASD. To date, studies of the brain and cognitive mechanisms that underlie this heterogeneity remain quite limited.

At the cognitive level, current research suggests that language impairment in verbal children with ASD involves deficits in phonological working memory, as evident on tests of nonsense word repetition. The areas of language that are most affected in this group include complex syntax and morphology related to marking tense (Tager-Flusberg et al., 2005). There is also considerable evidence from MRI (magnetic resonance imaging) studies of both children and adults that there are differences in volume and asymmetry in language regions of the cortex, specifically Broca's and Wernicke's areas. Recent studies suggest that these differences do not necessarily track with degree of language impairment, though there are conflicting findings in the literature. Importantly, most of the participants in cognitive and neuroimaging studies of ASD have been adults and individuals who have relatively intact language. Far less is known about the processes (either cognitive or neural) that might be implicated in the minimally verbal group. This project is designed to address this issue using two different brain imaging methods and approaches.

1. fMRI and DTI: Converging lines of evidence support the view that ASDs are disorders of connectivity, in which abnormalities in white matter integrity and reduced coordination of activity across brain regions give rise to core features. Recent results from our group (Guenther; Manoach) have identified white matter anomalies in the speech network of high-functioning verbal adults with ASD, specifically in the pathway between the left supplementary motor area (SMA) and left ventral premotor cortex (vPMC), a pathway involved in the initiation of speech output according to the Directions into Velocities of Articulators (DIVA) model of speech production, a leading model of the neural computations underlying speech. These connectivity abnormalities are revealed in both DTI and functional connectivity analyses collected using fMRI. NOTE: IRB approval for the collection of fMRI/DTI data will be obtained from MGH, where this portion of the study will be carried out. Data analyses will be carried out at MGH and BU.
2. Electrophysiology: EEG/ERP It has long been known that some children with ASD fail to respond when spoken to, cover their ears in the presence of certain sounds, yet show highly acute hearing in other contexts. Little is known about the mechanisms that might underlie these unusual auditory processing profiles. Abnormal neural oscillations have been found to be an endophenotype for ASD in infants and adults. However, the picture of how oscillations differ from those of non-clinical subjects is unclear and depends on the age at testing. Characterizing the oscillations present in the brains of a range of adolescents will allow us to quantify the relationship between neural activity and severity of language impairment. The main hypothesis that will be tested in this project is that abnormal neural connectivity in minimally verbal children with ASD profoundly impedes the ability to perceptually organize auditory scenes into meaningful units or objects, which has a direct effect on language development in these individuals. Event-related brain potentials (ERPs) and frequency-based analysis of the electroencephalogram (EEG) will be collected during passive listening tasks, to evaluate auditory perception and the perceptual organization of tones and speech using the mismatch negativity (MMN) paradigm (the MMN reflects passive deviance detection processes indexing low-level acoustic processes in automatic sensory memory mechanisms, and it has been widely investigated in studies of auditory perceptual discrimination of tones and speech).

The investigators plan to collect these data from 3 groups of adolescents with ASD varying in language skills (minimally verbal, verbal-language impaired, verbal-language normal) and age and gender matched non-ASD typical adolescents. The participants will be diagnosed and tested using a range of standardized and non-standardized assessments including IQ/cognitive level; social abilities; ASD severity; communication skills (nonverbal). These assessments will be carried out by trained examiners in the clinical core housed at BU.

Because many of the participants present with highly challenging behaviors and are difficult to test, a number of innovative approaches will be taken to maximize participants' success in completing the behavioral assessments, and then to tolerate and provide artifact-free data in the electrophysiological and MRI portions of the study.

Overall, the investigators hypothesize that the groups tested will differ in their neural indices of auditory perception, neural indices of perceptual organization, and induced neural oscillations. Further, the investigators hypothesize that differences in the degree of language impairment across these groups will be correlated with differences in the degree of abnormality of the measured neural indices, but not in the form of the abnormality, suggesting that the root causes of the differences across the tested subject groups are quantitative rather than qualitative.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14 and 21
* Minimally verbal (which is defined as having fewer than 10 words/phrases used communicatively during the Autism Diagnostic Observation Schedule (ADOS) assessment
* Demonstrated minimal progress in speech acquisition despite having participated in speech therapy for at least 18 months
* Diagnosis of Autism Spectrum Disorder (ASD)
* Verbal but language impaired (defined as more than 1.25 standard deviation below the mean on the clinical evaluation of language fundamentals - Fourth edition (CELF-4))
* Has normal language scores (on the CELF-4)
* Is typically developing with no history of psychiatric or neurological disorders

Exclusion Criteria:

* Has contraindications to having a magnetic resonance imaging (MRI) scan (e.g. electronic/ferromagnetic implant, clips, stents, existing or planned major dental work)
* Has a history of significant neurological diseases
* Has a history of sensory impairment (e.g., hearing impairment)
* Has a history of disorders other than ASD
* Is currently taking antipsychotic medications.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-02; Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Autism Spectrum Diagnosis | 5 years
  Interview
Adaptive Behaviors | 5 years
  Interview
Cognitive Abilities | 5 years
  Interview
Language Abilities | 5 years
  Interview and Questionnaire
Social Behavior | 5 years
  Interview
Repetitive Behavior | 5 years
  Questionnaire
Sensory Behavior | 5 years
  Questionnaire
Atypical Behavior | 5 years
  Questionnaire
Psychopathology | 5 years
  Questionnaire
Emotion Regulation | 5 years
  Questionnaire
Handedness | 5 years
  Questionnaire
Brain measures of structural and functional connectivity in key nodes of the speech production network | 5 years
  In particular between the supplementary motor area (SMA) and ventral premotor cortex (vPMC), a set of nodes in the speech network that is critical for the initiation of speech motor programs. High resolution MRI brain scans collected from adolescents with ASD who vary in their language ability from minimally verbal to normal (and a typical control group). Measures of structural anatomical connectivity based on Diffusion Tensor Imaging (DTI) data and functional connectivity based on resting state functional connectivity MRI.
Electrophysiological measures and neural oscillatory patterns of the perception, organization and analysis of auditory scenes. | 5 years
  Physiological parameter
Indices of social attention deployment measured by unobtrusively recording participants' eye-movements during the passive viewing of brief realistic video-clips. | 5 years
  Physiological parameter
Indices of electrodermal activity (EDA) measured wirelessly with the Q sensor (a small wearable device designed to work in real-world environments in an untethered, unobtrusive way). | 5 years
  Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Helen Tager-Flusberg, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tager-Flusberg H, Kasari C. Minimally verbal school-aged children with autism spectrum disorder: the neglected end of the spectrum. Autism Res. 2013 Dec;6(6):468-78. doi: 10.1002/aur.1329. Epub 2013 Oct 7. PMID 24124067
- See also: This is the website for our center. — http://www.bu.edu/autism